CLINICAL TRIAL: NCT01620255
Title: A Double-blind, Randomized, Placebo-controlled, Parallel, Dose-ranging Study To Evaluate The Efficacy And Safety Of Pf-00547659 In Subjects With Moderate To Severe Ulcerative Colitis (Turandot)
Brief Title: A Study Of PF-00547659 In Patients With Moderate To Severe Ulcerative Colitis
Acronym: TURANDOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A7281009; 2012-002030-37 (EudraCT Number); TURANDOT (Other: Alias Study Number)
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Drug Dose Level 1 (Experimental)
  Interventions: Drug: PF-00547659 SC Injection
- Drug Dose Level 2 (Experimental)
  Interventions: Drug: PF-00547659 SC Injection
- Drug Dose Level 3 (Experimental)
  Interventions: Drug: PF-00547659 SC Injection
- Drug Dose Level 4 (Experimental)
  Interventions: Drug: PF-00547659 SC Injection

INTERVENTIONS:
Drug: Placebo — Placebo delivered subcutaneous injection, 3 doses separated by 4 weeks
  Arms: Placebo
Drug: PF-00547659 SC Injection — Drug Dose Level 1 delivered subcutaneous injection, 3 doses separated by 4 weeks
  Arms: Drug Dose Level 1
Drug: PF-00547659 SC Injection — Drug Dose Level 2 delivered subcutaneous injection, 3 doses separated by 4 weeks
  Arms: Drug Dose Level 2
Drug: PF-00547659 SC Injection — Drug Dose Level 3 delivered subcutaneous injection, 3 doses separated by 4 weeks
  Arms: Drug Dose Level 3
Drug: PF-00547659 SC Injection — Drug Dose Level 4 delivered subcutaneous injection, 3 doses separated by 4 weeks
  Arms: Drug Dose Level 4

SUMMARY:
To determine the dose or doses of PF-00547659 that will be the most effective to improve or halt the disease symptoms in patients with moderate to severe ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis of Ulcerative Colitis for 3 or more months.
* Ulcerative colitis must be active beyond the rectum.
* Must active Ulcerative Colitis with a Total Mayo Score of 6 to 12 points

Exclusion Criteria:

* Pregnant or breast feeding.
* Diagnosis of indeterminate colitis or Crohn's Disease
* Subjects with history of colonic or small bowel obstruction or resection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2012-11-02 (Actual); Primary Completion 2014-09-22 (Actual); Study Completion 2016-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (190):
- United States (99):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - UCSD Health System-Pharmacy only, La Jolla, California
  - Clinical and Translational Research Institute, La Jolla, California
  - Perlman Medical Offices, La Jolla, California
  - Thornton Hospital, La Jolla, California
  - Community Clinical Trials, Orange, California
  - GastroDiagnostics - Community Clinical Trials Drug, Orange, California
  - Rocky Mountain Clinical Research, LLC., Denver, Colorado
  - Clinical Research of the Rockies, Lafayette, Colorado
  - Rocky Mountain Gastroenterology Associates, Thornton, Colorado
  - Endoscopy Center of Connecticut, LLC, Guilford, Connecticut
  - Endoscopy Center of Connecticut, LLC, Hamden, Connecticut
  - Gastroenterology Center of Connecticut, PC, Hamden, Connecticut
  - Medical REsearch Center of CT Drug, Hamden, Connecticut
  - Medical Research Network of Connecticut, Hamden, Connecticut
  - Florida Surgery Center, Altamonte Springs, Florida
  - Gastroenterology Associates, Crystal River, Florida
  - Research Consultant Group, Hialeah, Florida
  - Th Palmetto Surgery Center, Hialeah, Florida
  - Citrus Memorial Hospital, Inverness, Florida
  - Inverness Medical Imaging, Inverness, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Suncoast Endoscopy Center, Inverness, Florida
  - Sand Lake Imaging, Maitland, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Miami Hospital and Clinic - Local Lab, Miami, Florida
  - University of Miami Hospital and Clinic, Miami, Florida
  - University of Miami Hospital, Miami, Florida
  - Coral View Surgery Center, Miami, Florida
  - Center for Diagnostic Imaging, Miami Beach, Florida
  - First Quality Laboratory, Miramar, Florida
  - FQL Research, LLC, Miramar, Florida
  - Venutre Ambulatory Sugery Center, North Miami Beach, Florida
  - Boston Diagnostic Imaging, Orlando, Florida
  - Citrus Ambulatory Surgery Center, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Georgia Endoscopy Center, Alpharetta, Georgia
  - GI Consultants, Atlanta, Georgia
  - Atlanta Gastroenterology Specialist, Suwanee, Georgia
  - Covance Central Laboratory Services Inc, Indianapolis, Indiana
  - Covance Central Laboratory Services, Inc, Indianapolis, Indiana
  - Covance Laboratory Services, Inc, Indianapolis, Indiana
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Endoscopic Microsurgery Associates, Towson, Maryland
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Signature Healthcare Brockton, Brockton, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - East Valley Endoscopy, Grand Rapids, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Metro Health Endoscopy Unit, Wyoming, Michigan
  - Minneapolis Medical Eye Clinic, Minneapolis, Minnesota
  - Noran Neurology Clinic, Minneapolis, Minnesota
  - Minneapolis Heart Institute, Plymouth, Minnesota
  - Consulting Radiology, Plymouth, Minnesota
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Surgery Center of Columbia, Columbia, Missouri
  - Center for Digestive and Liver Diseases, Mexico, Missouri
  - Barnes-Jewish Hospital Investigational Drug Service (IP Shipping Address), St Louis, Missouri
  - Barnes-Jewish Hospital Radiology (X-Ray Only), St Louis, Missouri
  - Center for Advanced Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nevada School of Medicine (UNSOM), Las Vegas, Nevada
  - Las Vegas Surgery Center, Las Vegas, Nevada
  - Steinberg Diagnostic Medical Imaging Centers, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - New York Presbyterian Hospital - Weill Cornell Medical College, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College of Cornell University, New York, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - Premier Medical Group Research Department - Drug, Poughkeepsie, New York
  - UNC Hospitals Endoscopy Center At Meadowmont, Chapel Hill, North Carolina
  - Department of Pharmacy Investigational Drug Services, Chapel Hill, North Carolina
  - UNC Memorial Hospital, Chapel Hill, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Oregon Clinic, PC - Gastroenterology West, Portland, Oregon
  - Gastro One, Germantown, Tennessee
  - Diagnostic Imaging, Memphis, Tennessee
  - Vanderbilt University Medical Center: GI Clinical Research, Nashville, Tennessee
  - Vanderbilt University Medical Center: IBD Clinic, Nashville, Tennessee
  - Vanderbilt University Medical Center: Drug Shipment, Nashville, Tennessee
  - Vanderbilt University Medical Center: Endoscopy Lab, Nashville, Tennessee
  - Vanderbilt University Medical Center: Outpatient Radiology, Nashville, Tennessee
  - Houston Hospital for Specialized Surgery, Houston, Texas
  - Baylor Clinic (Drug Storage), Houston, Texas
  - Baylor College Of Medicine - Baylor Medical Center, Houston, Texas
  - Spring Gastroenterology and Associates, Humble, Texas
  - Spring Gastroenterology Drug, Humble, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Pioneer Research Solutions, Inc, Sugar Land, Texas
  - McGuire DVAMC, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - PI Radiology, Milwaukee, Wisconsin
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
  - Dynacare Laboratories, Wauwatosa, Wisconsin
  - GI associates drug, Wauwatosa, Wisconsin
- Australia (6):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Health Services, South Brisbane, Queensland
  - Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - The Canberra Hospital, Garran
- AKH Wien, Universitaetsklinik fuer Innere Medizin III, Vienna, Austria
- Belgium (3):
  - AZ St-Elisabeth Herentals, Herentals
  - University Hospital Gasthuisberg, Leuven
  - Centre Hospitalier de Mouscron, Mouscron
- Bulgaria (3):
  - 4- MBAL, Sofia
  - MBAL Sveti Ivan Rilski, Klinika po Gastroenterologia, Sofia
  - MBAL SofiaMed OOD, Sofia
- Canada (10):
  - GI Research Institute (GIRI), Vancouver, British Columbia
  - Office of Dr. David C. Pearson, Victoria, British Columbia
  - Office of Drs. Ranjit Andrew Singh and Jamie D. Papp, Victoria, British Columbia
  - PerCuro Clinical Research Limited, Victoria, British Columbia
  - Hamilton Health Sciences Corporation, McMaster University Medical Centre, Hamilton, Ontario
  - McMaster University Medical Center, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Oshawa Clinic, Oshawa, Ontario
  - Pavillion Rachel Tourigny, Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Czechia (3):
  - Hepato-Gastroenterology HK s.r.o., Hradec Králové
  - Klinické Centrum ISCARE I.V.F, Prague
  - Krajska zdravotni, a.s., Masarykova nemocnice v Usti nad Labem o.z., Ústí nad Labem
- France (7):
  - CHU Amiens - Hôpital Nord, Amiens
  - Centre Hospitalier Universitaire (CHU) de Caen - Hopital Cote de Nacre, Caen
  - Hopital Huriez CHRU de Lille, Lille
  - Hôpital l'Archet 2 CHU de Nice, Nice
  - Hopital Haut Leveque, Pessac
  - Hôpital Nord Service de Gastro-entérologie, Saint-Priest-en-Jarez
  - CHU Nancy - Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (3):
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitaetsklinik Regensburg, Regensburg
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart
- Hungary (2):
  - Pannonia Maganorvosi Centrum Kft, Budapest
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes
- Israel (5):
  - Digestive Disease Institute, Jerusalem
  - Gastroenterology and Liver Diseases Unit - Hadassah Ein Kerem University Hospital, Jerusalem
  - Dept. of Gastroenterology & Hepatology, Meir Medical Center, Kfar Saba
  - Gastroenterology Division, Rabin Medical Center, Beilinson Campus, Petah Tikva
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (9):
  - Universita' degli Studi "Magna Graecia" di Catanzaro, UO di Fisiopatologia Digestiva, Catanzaro
  - IBD Center - Divisione Gastroenterologia - Istituto Clinico Humanitas IRCCS, Milan
  - IRCCS Policlinico San Donato, Milan
  - Azienda Ospedaliera -Università di Padova, Padua
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Azienda Ospedaliera Universitaria, Policlinico Tor Vergata, Roma
  - Universita Cattolica Sacro Cuore Policlinico "A. Gemelli", Roma
  - AOS San Camillo Forlanini, Rome
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Netherlands (3):
  - Academic Medical Center - University of Amsterdam, Amsterdam, North Holland
  - University Medical Center Groningen (UMCG), Groningen
  - Maastricht University Medical Center, Maastricht
- New Zealand (6):
  - Christchurch Hospital, Christchurch
  - Southern Endoscopy Centre, Christchurch
  - Midland Neurology & EMG Ltd., Hamilton
  - The Hamilton Eye Clinic, Hamilton
  - Cardiac Services Ltd., Hamilton
  - Waikato Hospital, Hamilton
- Poland (8):
  - Centrum endoskopii Zabiegowej, Poradnia Chorob Jelitowych,, Bydgoszcz
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Centrum Medyczne - Szpital Swietej Rodziny Sp. z o.o., Lodz
  - Centrum Medyczne HCP Lecznictwo Ambulatoryjne Pracownia Endoskopowa, Poznan
  - Klinika Chorob Wewnetrznych i Gastroenterologii z Pododdzialem, Warsaw
  - NZOZ Vivamed, Warsaw
  - Wojskowy Szpital Kliniczny z Poliklinika SPOZ, Wroclaw
  - Lexmedica, Wroclaw
- SBEI of HPE North-West State Medical University n.a. I.I. Mechnikov of the MH of the RF St.P SBIH ", Saint Petersburg, Russia
- Serbia (5):
  - Clinical Hospital Centre Bezanijska Kosa, Clinic for Internal medicine, Belgrade
  - Clinical Hospital Centre Zvezdara Clinic for Gastroenterology and Hepatology, Belgrade
  - Military medical Academy, Belgrade
  - Clinical Hospital Center Zemun, Gastroenterology and Hepatology Department, Belgrade
  - Clinical Centre of Nis, Clinic for Gastroenterology and Hepatology, Niš
- Slovakia (4):
  - Gastro I., s.r.o., Prešov, Slovak Republic
  - Gastroenterological Centre Thalion, Bratislava
  - KM Management spol. s.r.o. Gastroenterologicke a hepatologicke centrum Nitra, Nitra
  - Ustredna vojenska nemocnice SNP Ruzomberok, Ružomberok
- Kingsbury Hospital, Claremont, CAPE TOWN, South Africa
- South Korea (7):
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei University College of Medicine, Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Parc de Salut Mar-Hospital del Mar, Barcelona
  - Centro Medico Teknon, Barcelona
  - Hospital Clinic de Barcelona, Barcelona

REFERENCES:
- [Derived] Zhou H, Xi L, Ziemek D, O'Neil S, Lee J, Stewart Z, Zhan Y, Zhao S, Zhang Y, Page K, Huang A, Maciejewski M, Zhang B, Gorelick KJ, Fitz L, Pradhan V, Cataldi F, Vincent M, Von Schack D, Hung K, Hassan-Zahraee M. Molecular Profiling of Ulcerative Colitis Subjects from the TURANDOT Trial Reveals Novel Pharmacodynamic/Efficacy Biomarkers. J Crohns Colitis. 2019 May 27;13(6):702-713. doi: 10.1093/ecco-jcc/jjy217. PMID 30901380
- [Derived] Vermeire S, Sandborn WJ, Danese S, Hebuterne X, Salzberg BA, Klopocka M, Tarabar D, Vanasek T, Gregus M, Hellstern PA, Kim JS, Sparrow MP, Gorelick KJ, Hinz M, Ahmad A, Pradhan V, Hassan-Zahraee M, Clare R, Cataldi F, Reinisch W. Anti-MAdCAM antibody (PF-00547659) for ulcerative colitis (TURANDOT): a phase 2, randomised, double-blind, placebo-controlled trial. Lancet. 2017 Jul 8;390(10090):135-144. doi: 10.1016/S0140-6736(17)30930-3. Epub 2017 May 17. PMID 28527704
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7281009&StudyName=A%20study%20Of%20PF-00547659%20In%20Patients%20With%20Moderate%20To%20Severe%20Ulcerative%20Colitis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two (2) subjects initially randomized to the 22.5 mg group were mistakenly administered the 75 mg dose instead and were counted under that group. The numbers Started reflect the number of participants who received treatment.
Groups:
- Placebo: Participants received placebo in the form of 3 subcutaneous (SC) injections on Days 1, 28, and 56, following the completion of most study procedures. Participants were administered placebo SC in the anterolateral right or left thighs. Injections were administered at least 3 centimeters (cm) apart to the same thigh beginning from the outermost section of the thigh OR 2 injections in 1 thigh about 3 cm apart and 1 in the other thigh.
- PF-00547659 7.5 mg: Participants received PF-00547659 7.5 milligrams (mg) in the form of 3 subcutaneous (SC) injections on Days 1, 28, and 56, following the completion of most study procedures. Participants were administered PF-00547659 7.5 mg SC in the anterolateral right or left thighs. Injections were administered at least 3 cm apart to the same thigh beginning from the outermost section of the thigh OR 2 injections in 1 thigh about 3 cm apart and 1 in the other thigh.
- PF-00547659 22.5 mg: Participants received PF-00547659 22.5 milligrams (mg) in the form of 3 subcutaneous (SC) injections on Days 1, 28, and 56, following the completion of most study procedures. Participants were administered PF-00547659 22.5 mg SC in the anterolateral right or left thighs. Injections were administered at least 3 cm apart to the same thigh beginning from the outermost section of the thigh OR 2 injections in 1 thigh about 3 cm apart and 1 in the other thigh.
- PF-00547659 75 mg: Participants received PF-00547659 75 milligrams (mg) in the form of 3 subcutaneous (SC) injections on Days 1, 28, and 56, following the completion of most study procedures. Participants were administered PF-00547659 75 mg SC in the anterolateral right or left thighs. Injections were administered at least 3 cm apart to the same thigh beginning from the outermost section of the thigh OR 2 injections in 1 thigh about 3 cm apart and 1 in the other thigh.
- PF-00547659 225 mg: Participants received PF-00547659 225 milligrams (mg) in the form of 3 subcutaneous (SC) injections on Days 1, 28, and 56, following the completion of most study procedures. Participants were administered PF-00547659 225 mg SC in the anterolateral right or left thighs. Injections were administered at least 3 cm apart to the same thigh beginning from the outermost section of the thigh OR 2 injections in 1 thigh about 3 cm apart and 1 in the other thigh.
Period: Overall Study
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Started | 73 | 71 | 70 | 73 | 70
Treated | 73 | 71 | 70 | 73 | 70
Completed | 69 | 65 | 68 | 70 | 64
Not Completed | 4 | 6 | 2 | 3 | 6
Not completed — Withdrawal by Subject | 4 | 1 | 1 | 2 | 4
Not completed — Participant underwent fecal transplant | 0 | 0 | 1 | 0 | 0
Not completed — Non-compliance | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 4 | 0 | 1 | 1
Not completed — Withdrawn at discretion of investigator | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo in the form of 3 subcutaneous (SC) injections on Days 1, 28, and 56, following the completion of most study procedures. Participants were administered placebo SC in the anterolateral right or left thighs. Injections were administered at least 3 cm apart to the same thigh beginning from the outermost section of the thigh OR 2 injections in 1 thigh about 3 cm apart and 1 in the other thigh.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg | Total
Number analyzed (Participants) | 73 | 71 | 70 | 73 | 70 | 357
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (12.7) | 41.3 (12.5) | 42.1 (14.7) | 37.7 (12.4) | 41.3 (13.2) | 40.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 25 | 35 | 28 | 149
  Male | 44 | 39 | 45 | 38 | 42 | 208

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Clinical Remission at Week 12
Description: Clinical remission was defined as a Total Mayo Score of less than or equal (<=) 2 points with no individual subscore exceeding 1 point and rectal bleed subscore of 0 or 1. The Mayo Score is a tool designed to measure disease activity for ulcerative colitis (UC). Scoring ranges from 0 to 12 points and consists of 4 subscores, each graded 0 to 3 with higher score indicating more severe disease activity. Endoscopic readings from the local and the central reader were considered for analysis. The central reading was used as the primary analysis and the local readings were used for the sensitivity analyses.
Time Frame: Week 12
Population: The primary analysis population was based on a modified intent-to-treat (mITT) analysis set, which was defined as all randomized participants who received at least 1 dose of randomized treatment. Two subjects initially randomized to the 22.5 mg group were mistakenly administered the 75 mg dose instead.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 73 | 71 | 72 | 71 | 70
percentage of participants
  Centrally read | 2.7 [0.7 to 7.6] | 11.3 [5.7 to 18.8] | 16.7 [9.9 to 25.4] | 15.5 [9.5 to 23.6] | 5.7 [2.5 to 12.5]
  Locally read | 5.5 [2.4 to 12.0] | 14.1 [7.8 to 22.0] | 23.6 [15.6 to 33.1] | 18.3 [11.9 to 27.1] | 12.9 [7.3 to 21.1]
Statistical Analysis 1: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg versus (vs) placebo, centrally read; Test type: Superiority or Other; p = 0.0213, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.080, 90% CI 2-sided [0.019 to 0.140] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 2: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, centrally read; Test type: Superiority or Other; p = 0.0025, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.128, 90% CI 2-sided [0.056 to 0.199] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 3: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, centrally read; Test type: Superiority or Other; p = 0.0040, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.118, 90% CI 2-sided [0.048 to 0.188] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 4: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, centrally read; Test type: Superiority or Other; p = 0.1803, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.026, 90% CI 2-sided [-0.012 to 0.064] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 5: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.0582, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.080, 90% CI 2-sided [0.002 to 0.159] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 6: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.0014, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.178, 90% CI 2-sided [0.083 to 0.272] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 7: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.0125, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.122, 90% CI 2-sided [0.036 to 0.208] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 8: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.0927, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.066, 90% CI 2-sided [-0.009 to 0.142] — Statistics of risk difference are calculated using the Minimum Risk Weights test

2. Secondary Outcome: Percentage of Participants With Clinical Response at Week 12
Description: Clinical response was defined as a decrease from baseline of at least 3 points in Total Mayo Score with at least a 30 percent (%) change, accompanied by at least 1 point decrease or absolute score of 0 or 1 in rectal bleeding subscore. The Mayo Score is a tool designed to measure disease activity for UC. Scoring ranges from 0 to 12 points and consists of 4 subscores, each graded 0 to 3 with higher score indicating more severe disease activity. Endoscopic readings from the local and the central reader were considered for analysis. The central reading was used as the primary analysis and the local readings were used for the sensitivity analyses.
Time Frame: Week 12
Population: The primary analysis population was based on an mITT analysis set, which was defined as all randomized participants who received at least 1 dose of randomized treatment. n=number of participants evaluable for the specified category.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 73 | 71 | 72 | 71 | 70
percentage of participants
  Centrally read (n=73,71,72,71,70) | 28.8 [20.2 to 37.8] | 38.0 [28.4 to 47.6] | 54.2 [44.2 to 64.2] | 45.1 [35.0 to 55.3] | 50.0 [39.6 to 60.4]
  Locally read (n=73,70,72,70,70) | 32.9 [24.2 to 42.3] | 38.6 [28.8 to 48.1] | 54.2 [44.2 to 64.2] | 48.6 [38.2 to 59.0] | 51.4 [41.0 to 61.8]
Statistical Analysis 1: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, centrally read; Test type: Superiority or Other; p = 0.1379, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.089, 90% CI 2-sided [-0.037 to 0.214] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 2: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, centrally read; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.254, 90% CI 2-sided [0.121 to 0.388] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 3: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, centrally read; Test type: Superiority or Other; p = 0.0239, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.163, 90% CI 2-sided [0.032 to 0.293] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 4: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, centrally read; Test type: Superiority or Other; p = 0.0052, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.213, 90% CI 2-sided [0.080 to 0.347] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 5: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.2617, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.056, 90% CI 2-sided [-0.075 to 0.186] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 6: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.0058, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.212, 90% CI 2-sided [0.077 to 0.347] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 7: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.0326, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.156, 90% CI 2-sided [0.022 to 0.290] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 8: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.0145, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.185, 90% CI 2-sided [0.050 to 0.320] — Statistics of risk difference are calculated using the Minimum Risk Weights test

3. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 12
Description: Mucosal healing was defined as absolute Mayo subscore for endoscopy of 0 or 1. The Mayo Score is a tool designed to measure disease activity for UC. Scoring ranges from 0 to 12 points and consists of 4 subscores, each graded 0 to 3 with higher score indicating more severe disease activity. Endoscopic readings from the local and the central reader were considered for analysis. The central reading was used as the primary analysis and the local readings were used for the sensitivity analyses.
Time Frame: Week 12
Population: The primary analysis population was based on an mITT analysis set, which was defined as all randomized participants who received at least 1 dose of randomized treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 73 | 71 | 72 | 71 | 70
percentage of participants
  Centrally read | 8.2 [3.6 to 15.4] | 15.5 [9.5 to 23.6] | 27.8 [19.5 to 37.1] | 25.4 [17.1 to 35.0] | 14.3 [8.0 to 22.3]
  Locally read | 21.9 [14.9 to 31.4] | 22.5 [15.4 to 31.6] | 37.5 [28.0 to 47.2] | 35.2 [25.8 to 44.7] | 28.6 [20.2 to 38.2]
Statistical Analysis 1: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, centrally read; Test type: Superiority or Other; p = 0.0618, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.081, 90% CI 2-sided [0.000 to 0.162] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 2: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, centrally read; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.187, 90% CI 2-sided [0.091 to 0.284] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 3: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, centrally read; Test type: Superiority or Other; p = 0.0027, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.159, 90% CI 2-sided [0.068 to 0.250] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 4: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, centrally read; Test type: Superiority or Other; p = 0.0999, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.069, 90% CI 2-sided [-0.013 to 0.151] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 5: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.5225, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.001, 90% CI 2-sided [-0.111 to 0.114] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 6: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.0246, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.154, 90% CI 2-sided [0.030 to 0.278] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 7: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.0464, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.130, 90% CI 2-sided [0.008 to 0.253] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 8: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, locally read; Test type: Superiority or Other; p = 0.2000, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.066, 90% CI 2-sided [-0.053 to 0.186] — Statistics of risk difference are calculated using the Minimum Risk Weights test

4. Secondary Outcome: Percentage of Participants With Absolute Partial Mayo Score of Less Than or Equal to (<=) 2 With no Individual Subscore More Than (>) 1 at Weeks 4, 8, and 12
Description: An absolute Partial Mayo Score of <=2 corresponds to remission. However, this endpoint was incorrectly stated in the protocol and instead of "absolute Partial Mayo Score <=2", it was stated as "change from baseline in Partial Mayo Score <=2".
Time Frame: Weeks 4, 8, and 12
Population: As this endpoint was incorrectly stated in the protocol, no analyses were done and no data are presented.
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Total Mayo Score at Week 12
Description: The Mayo Score is a tool designed to measure disease activity for UC. Scoring ranges from 0 to 12 points and consists of 4 subscores, each graded 0 to 3 with higher score indicating more severe disease activity. Endoscopic readings from the local and the central reader were considered for analysis. The central reading was used as the primary analysis and the local readings were used for the sensitivity analyses.
Time Frame: Baseline, Week 12
Population: The primary analysis population was based on an mITT analysis set, which was defined as all randomized participants who received at least 1 dose of randomized treatment. n=number of evaluable participants in that specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 73 | 71 | 72 | 71 | 70
units on a scale
  Centrally read baseline (n=73,71,72,71,70) | 8.4 (1.71) | 8.7 (1.65) | 8.1 (1.63) | 8.4 (1.94) | 8.7 (1.60)
  Centrally read change (n=67,63,69,67,63) | -1.5 (2.42) [-2.043 to -1.014] | -2.4 (2.78) [-2.944 to -1.881] | -2.9 (2.49) [-3.570 to -2.550] | -2.5 (2.74) [-3.162 to -2.131] | -2.9 (2.78) [-3.337 to -2.270]
  Locally read baseline (n=73,70,72,70,70) | 8.4 (1.72) | 8.8 (1.59) | 8.1 (1.72) | 8.3 (1.99) | 8.6 (1.62)
  Locally read change (n=67,62,70,66,64) | -1.7 (2.55) [-2.280 to -1.171] | -2.7 (3.05) [-3.241 to -2.084] | -3.1 (2.70) [-3.866 to -2.775] | -2.7 (2.92) [-3.357 to -2.236] | -3.1 (3.07) [-3.583 to -2.442]
Statistical Analysis 1: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, centrally read change; Test type: Superiority or Other; p = 0.0494, ANCOVA; Analysis of covariance (ANCOVA) with model terms: treatment group, baseline, status of anti-tumor necrosis factor (TNF) therapy experience; Least Squares Mean (LSM) Difference = -0.88, 90% CI 2-sided [-1.623 to -0.145]
Statistical Analysis 2: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, centrally read change; Test type: Superiority or Other; p = 0.0005, ANCOVA; [statistical method as in outcome 5, analysis 1]; LSM Difference = -1.53, 90% CI 2-sided [-2.254 to -0.809]
Statistical Analysis 3: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, centrally read change; Test type: Superiority or Other; p = 0.0117, ANCOVA; [statistical method as in outcome 5, analysis 1]; LSM Difference = -1.12, 90% CI 2-sided [-1.845 to -0.390]
Statistical Analysis 4: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, centrally read change; Test type: Superiority or Other; p = 0.0049, ANCOVA; [statistical method as in outcome 5, analysis 1]; LSM Difference = -1.27, 90% CI 2-sided [-2.016 to -0.533]
Statistical Analysis 5: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, locally read change; Test type: Superiority or Other; p = 0.0543, ANCOVA; [statistical method as in outcome 5, analysis 1]; LSM Difference = -0.94, 90% CI 2-sided [-1.737 to -0.137]
Statistical Analysis 6: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, locally read change; Test type: Superiority or Other; p = 0.0008, ANCOVA; [statistical method as in outcome 5, analysis 1]; LSM Difference = -1.60, 90% CI 2-sided [-2.372 to -0.819]
Statistical Analysis 7: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, locally read change; Test type: Superiority or Other; p = 0.0255, ANCOVA; [statistical method as in outcome 5, analysis 1]; LSM Difference = -1.07, 90% CI 2-sided [-1.858 to -0.284]
Statistical Analysis 8: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, locally read change; Test type: Superiority or Other; p = 0.0079, ANCOVA; [statistical method as in outcome 5, analysis 1]; LSM Difference = -1.29, 90% CI 2-sided [-2.082 to -0.493]

6. Secondary Outcome: Percentage of Participants With Change From Baseline in Individual Mayo Subscores - Stool Frequency, Rectal Bleeding, and Physician's Global Assessment (PGA) - at Weeks 4, 8, and 12
Description: The Mayo Score is a tool designed to measure disease activity for UC. Scoring ranges from 0 to 12 points and consists of 4 subscores (stool frequency, rectal bleeding, PGA, findings on flexible sigmoidoscopy), each graded 0 to 3 with higher score indicating more severe disease activity. Endoscopic readings from the local and the central reader were considered for analysis. The central reading was used as the primary analysis and the local readings were used for the sensitivity analyses. Changes from baseline in the subscore of less than (<) 0, 0, and >0 corresponded to improvement (imp), no change (NC), and worsening (wors) in that specific subscore.
Time Frame: Baseline; Weeks (W) 4, 8, and 12
Population: The primary analysis population was based on an mITT analysis set, which was defined as all randomized participants who received at least 1 dose of randomized treatment. n=number of evaluable participants at that specific time point for that endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 73 | 71 | 72 | 71 | 70
percentage of participants
  Imp in Stool frequency, W4 (n=67,64,71,69,65) | 26.87 [-2.043 to -1.014] | 46.88 [-2.944 to -1.881] | 36.62 [-3.570 to -2.550] | 30.43 [-3.162 to -2.131] | 43.08 [-3.337 to -2.270]
  NC in Stool frequency, W4 (n=67,64,71,69,65) | 59.70 [-2.280 to -1.171] | 42.19 [-3.241 to -2.084] | 60.56 [-3.866 to -2.775] | 63.77 [-3.357 to -2.236] | 52.31 [-3.583 to -2.442]
  Wors in Stool frequency, W4 (n=67,64,71,69,65) | 13.43 | 10.94 | 2.82 | 5.80 | 4.62
  Imp in Stool frequency, W8 (n=71,63,71,69,68) | 28.17 | 49.21 | 43.66 | 49.28 | 51.47
  NC in Stool frequency, W8 (n=71,63,71,69,68) | 60.56 | 42.86 | 53.52 | 46.38 | 48.53
  Wors in Stool frequency, W8 (n=71,63,71,69,68) | 11.27 | 7.94 | 2.82 | 4.35 | 0
  Imp in Stool frequency, W12 (n=67,63,71,68,64) | 35.82 | 49.21 | 56.34 | 45.59 | 56.25
  NC in Stool frequency, W12 (n=67,63,71,68,64) | 52.24 | 41.27 | 38.03 | 48.53 | 37.50
  Wors in Stool frequency, W12 (n=67,63,71,68,64) | 11.94 | 9.52 | 5.63 | 5.88 | 6.25
  Imp in Rectal Bleeding, W4 (n=67,64,71,69,65) | 22.39 | 48.44 | 42.25 | 42.03 | 49.23
  NC in Rectal Bleeding, W4 (n=67,64,71,69,65) | 62.69 | 42.19 | 57.75 | 53.62 | 44.62
  Wors in Rectal Bleeding, W4 (n=67,64,71,69,65) | 14.93 | 9.38 | 0 | 4.35 | 6.15
  Imp in Rectal Bleeding, W8 (n=71,63,71,69,68) | 33.80 | 50.79 | 40.85 | 46.38 | 64.71
  NC in Rectal Bleeding, W8 (n=71,63,71,69,68) | 54.93 | 36.51 | 50.70 | 44.93 | 33.82
  Wors in Rectal Bleeding, W8 (n=71,63,71,69,68) | 11.27 | 12.70 | 8.45 | 8.70 | 1.47
  Imp in Rectal Bleeding, W12 (n=67,63,71,68,64) | 37.31 | 53.97 | 50.70 | 47.06 | 60.94
  NC in Rectal Bleeding, W12 (n=67,63,71,68,64) | 50.75 | 34.92 | 42.25 | 45.59 | 35.94
  Wors in Rectal Bleeding, W12 (n=67,63,71,68,64) | 11.94 | 11.11 | 7.04 | 7.35 | 3.13
  Imp in PGA, W4 (n=67,64,71,69,65) | 47.76 | 57.81 | 56.34 | 56.52 | 60.00
  NC in PGA, W4 (n=67,64,71,69,65) | 49.25 | 34.38 | 39.44 | 42.03 | 35.38
  Wors in PGA, W4 (n=67,64,71,69,65) | 2.99 | 7.81 | 4.23 | 1.45 | 4.62
  Imp in PGA, W8 (n=71,63,71,69,68) | 59.15 | 61.90 | 66.20 | 62.32 | 67.65
  NC in PGA, W8 (n=71,63,71,69,68) | 33.80 | 30.16 | 30.99 | 37.68 | 30.88
  Wors in PGA, W8 (n=71,63,71,69,68) | 7.04 | 7.94 | 2.82 | 0 | 1.47
  Imp in PGA, W12 (n=67,63,71,68,64) | 50.75 | 61.90 | 64.79 | 55.88 | 57.81
  NC in PGA, W12 (n=67,63,71,68,64) | 43.28 | 31.75 | 32.39 | 39.71 | 32.81
  Wors in PGA, W12 (n=67,63,71,68,64) | 5.97 | 6.35 | 2.82 | 4.41 | 9.38
Statistical Analysis 1: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Stool Frequency, W4; Test type: Superiority or Other; p = 0.1016, Mixed Models Analysis; Linear Mixed Model (LMM) with model terms: treatment group, time, baseline, time by treatment, status of previous anti-TNF therapy experience; LSM Difference = -0.25, 90% CI 2-sided [-0.511 to 0.001]
Statistical Analysis 2: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Stool Frequency, W4; Test type: Superiority or Other; p = 0.0654, Mixed Models Analysis; LMM with model terms: treatment group, time, baseline, time by treatment, status of previous anti-TNF therapy experience; LSM Difference = -0.28, 90% CI 2-sided [-0.529 to -0.030]
Statistical Analysis 3: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, Stool Frequency, W4; Test type: Superiority or Other; p = 0.1500, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.22, 90% CI 2-sided [-0.472 to 0.031]
Statistical Analysis 4: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Stool Frequency, W4; Test type: Superiority or Other; p = 0.0132, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.38, 90% CI 2-sided [-0.637 to -0.129]
Statistical Analysis 5: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Stool Frequency, W8; Test type: Superiority or Other; p = 0.0526, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.30, 90% CI 2-sided [-0.555 to -0.046]
Statistical Analysis 6: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Stool Frequency, W8; Test type: Superiority or Other; p = 0.0422, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.31, 90% CI 2-sided [-0.554 to -0.058]
Statistical Analysis 7: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, Stool Frequency, W8; Test type: Superiority or Other; p = 0.0110, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.39, 90% CI 2-sided [-0.637 to -0.137]
Statistical Analysis 8: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Stool Frequency, W8; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.50, 90% CI 2-sided [-0.755 to -0.254]
Statistical Analysis 9: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Stool Frequency, W12; Test type: Superiority or Other; p = 0.1611, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.22, 90% CI 2-sided [-0.475 to 0.038]
Statistical Analysis 10: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Stool Frequency, W12; Test type: Superiority or Other; p = 0.0186, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.36, 90% CI 2-sided [-0.608 to -0.108]
Statistical Analysis 11: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, Stool Frequency, W12; Test type: Superiority or Other; p = 0.1647, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.21, 90% CI 2-sided [-0.465 to 0.039]
Statistical Analysis 12: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Stool Frequency, W12; Test type: Superiority or Other; p = 0.0231, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.35, 90% CI 2-sided [-0.607 to -0.097]
Statistical Analysis 13: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Rectal Bleeding, W4; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.46, 90% CI 2-sided [-0.658 to -0.260]
Statistical Analysis 14: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Rectal Bleeding, W4; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.52, 90% CI 2-sided [-0.710 to -0.322]
Statistical Analysis 15: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, Rectal Bleeding, W4; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.49, 90% CI 2-sided [-0.686 to -0.295]
Statistical Analysis 16: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Rectal Bleeding, W4; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.39, 90% CI 2-sided [-0.587 to -0.192]
Statistical Analysis 17: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Rectal Bleeding, W8; Test type: Superiority or Other; p = 0.0207, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.28, 90% CI 2-sided [-0.475 to -0.081]
Statistical Analysis 18: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Rectal Bleeding, W8; Test type: Superiority or Other; p = 0.0402, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.24, 90% CI 2-sided [-0.432 to -0.048]
Statistical Analysis 19: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, Rectal Bleeding, W8; Test type: Superiority or Other; p = 0.0071, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.32, 90% CI 2-sided [-0.511 to -0.124]
Statistical Analysis 20: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Rectal Bleeding, W8; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.47, 90% CI 2-sided [-0.664 to -0.275]
Statistical Analysis 21: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Rectal Bleeding, W12; Test type: Superiority or Other; p = 0.0395, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.25, 90% CI 2-sided [-0.449 to -0.050]
Statistical Analysis 22: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Rectal Bleeding, W12; Test type: Superiority or Other; p = 0.0073, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.32, 90% CI 2-sided [-0.511 to -0.123]
Statistical Analysis 23: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, Rectal Bleeding, W12; Test type: Superiority or Other; p = 0.0413, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.24, 90% CI 2-sided [-0.439 to -0.047]
Statistical Analysis 24: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Rectal Bleeding, W12; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.40, 90% CI 2-sided [-0.602 to -0.206]
Statistical Analysis 25: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, PGA, W4; Test type: Superiority or Other; p = 0.1862, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.19, 90% CI 2-sided [-0.421 to 0.046]
Statistical Analysis 26: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, PGA, W4; Test type: Superiority or Other; p = 0.0998, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.23, 90% CI 2-sided [-0.455 to -0.000]
Statistical Analysis 27: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, PGA, W4; Test type: Superiority or Other; p = 0.1085, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.22, 90% CI 2-sided [-0.453 to 0.006]
Statistical Analysis 28: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, PGA, W4; Test type: Superiority or Other; p = 0.3161, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.14, 90% CI 2-sided [-0.372 to 0.090]
Statistical Analysis 29: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, PGA, W8; Test type: Superiority or Other; p = 0.4962, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.10, 90% CI 2-sided [-0.328 to 0.136]
Statistical Analysis 30: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, PGA, W8; Test type: Superiority or Other; p = 0.0371, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.29, 90% CI 2-sided [-0.512 to -0.060]
Statistical Analysis 31: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, PGA, W8; Test type: Superiority or Other; p = 0.1212, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.21, 90% CI 2-sided [-0.441 to 0.013]
Statistical Analysis 32: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, PGA, W8; Test type: Superiority or Other; p = 0.1870, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.18, 90% CI 2-sided [-0.410 to 0.045]
Statistical Analysis 33: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, PGA, W12; Test type: Superiority or Other; p = 0.1133, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.23, 90% CI 2-sided [-0.459 to 0.009]
Statistical Analysis 34: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, PGA, W12; Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.43, 90% CI 2-sided [-0.653 to -0.198]
Statistical Analysis 35: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, PGA, W12; Test type: Superiority or Other; p = 0.0788, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.25, 90% CI 2-sided [-0.475 to -0.016]
Statistical Analysis 36: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, PGA, W12; Test type: Superiority or Other; p = 0.0717, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.25, 90% CI 2-sided [-0.485 to -0.022]

7. Secondary Outcome: Percentage of Participants With Change From Baseline in Individual Mayo Subscore - Findings on Flexible Sigmoidoscopy - at Week 12
Description: The Mayo Score is a tool designed to measure disease activity for UC. Scoring ranges from 0 to 12 points and consists of 4 subscores (stool frequency, rectal bleeding, PGA, findings on flexible sigmoidoscopy), each graded 0 to 3 with higher score indicating more severe disease activity. Endoscopic readings from the local and the central reader were considered for analysis. The central reading was used as the primary analysis and the local readings were used for the sensitivity analyses. Changes from baseline in the subscore of <0, 0, and >0 corresponded to improvement (imp), no change (NC), and worsening (wors) in that specific subscore.
Time Frame: Baseline, Week 12
Population: The primary analysis population was based on an mITT analysis set, which was defined as all randomized participants who received at least 1 dose of randomized treatment. n=number of evaluable participants at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 73 | 71 | 72 | 71 | 70
percentage of participants
  Imp (n=67,63,69,67,63) | 25.37 [-2.043 to -1.014] | 28.57 [-2.944 to -1.881] | 47.83 [-3.570 to -2.550] | 47.76 [-3.162 to -2.131] | 39.68 [-3.337 to -2.270]
  NC (n=67,63,69,67,63) | 61.19 [-2.280 to -1.171] | 60.32 [-3.241 to -2.084] | 49.28 [-3.866 to -2.775] | 46.27 [-3.357 to -2.236] | 57.14 [-3.583 to -2.442]
  Wors (n=67,63,69,67,63) | 13.43 | 11.11 | 2.90 | 5.97 | 3.17
Statistical Analysis 1: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo; Test type: Superiority or Other; p = 0.5406, ANCOVA; ANCOVA with model terms: treatment group, baseline, status of anti-TNF therapy experience; LSM Difference = -0.08, 90% CI 2-sided [-0.286 to 0.131]
Statistical Analysis 2: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo; Test type: Superiority or Other; p = 0.0007, ANCOVA; ANCOVA with model terms: treatment group, baseline, status of anti-TNF therapy experience; LSM Difference = -0.42, 90% CI 2-sided [-0.628 to -0.221]
Statistical Analysis 3: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo; Test type: Superiority or Other; p = 0.0063, ANCOVA; ANCOVA with model terms: treatment group, baseline, status of anti-TNF therapy experience; LSM Difference = -0.34, 90% CI 2-sided [-0.549 to -0.137]
Statistical Analysis 4: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo; Test type: Superiority or Other; p = 0.0748, ANCOVA; ANCOVA with model terms: treatment group, baseline, status of anti-TNF therapy experience; LSM Difference = -0.23, 90% CI 2-sided [-0.436 to -0.018]

8. Secondary Outcome: Percent Change From Baseline in Fecal Calprotectin at Weeks 4, 8, and 12
Description: Fecal calprotectin was one of the pharmacodynamic (PD) biomarkers of the study.
Time Frame: Baseline, Weeks 4, 8, and 12
Population: The primary analysis population was based on an mITT analysis set, which was defined as all randomized participants who received at least 1 dose of randomized treatment. n=number of evaluable participants at that specific time point.
Measure: Geometric Mean (90% Confidence Interval); unit: percent change
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 73 | 71 | 72 | 71 | 70
percent change
  Week 4 (n=62,57,68,67,60) | -25.62 [-43.49 to -2.09] | -40.21 [-55.56 to -19.54] | -23.50 [-44.27 to 5.00] | -46.22 [-61.46 to -24.95] | -39.27 [-56.74 to -14.75]
  Week 8 (n=67,57,67,63,65) | -21.68 [-39.62 to 1.60] | -44.49 [-60.05 to -22.88] | -44.77 [-60.49 to -22.80] | -57.20 [-69.74 to -39.45] | -49.54 [-65.08 to -27.07]
  Week 12 (n=61,55,64,64,59) | -22.59 [-42.68 to 4.54] | -56.34 [-69.39 to -37.72] | -58.41 [-72.26 to -37.65] | -56.72 [-71.67 to -33.88] | -64.52 [-76.92 to -45.43]
Statistical Analysis 1: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Week 4; Test type: Superiority or Other; p = 0.9744, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -1.9, 90% CI 2-sided [-101.00 to 97.14]
Statistical Analysis 2: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Week 4; Test type: Superiority or Other; p = 0.2023, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 74.9, 90% CI 2-sided [-21.77 to 171.66]
Statistical Analysis 3: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, Week 4; Test type: Superiority or Other; p = 0.5808, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 32.9, 90% CI 2-sided [-65.09 to 130.79]
Statistical Analysis 4: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Week 4; Test type: Superiority or Other; p = 0.5388, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 37.6, 90% CI 2-sided [-63.12 to 138.34]
Statistical Analysis 5: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Week 8; Test type: Superiority or Other; p = 0.8902, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -8.2, 90% CI 2-sided [-106.24 to 89.81]
Statistical Analysis 6: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Week 8; Test type: Superiority or Other; p = 0.8616, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 10.2, 90% CI 2-sided [-86.14 to 106.54]
Statistical Analysis 7: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, Week 8; Test type: Superiority or Other; p = 0.5684, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -34.3, 90% CI 2-sided [-133.49 to 64.79]
Statistical Analysis 8: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Week 8; Test type: Superiority or Other; p = 0.5700, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 33.8, 90% CI 2-sided [-64.20 to 131.86]
Statistical Analysis 9: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Week 12; Test type: Superiority or Other; p = 0.6234, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -30.0, 90% CI 2-sided [-130.56 to 70.57]
Statistical Analysis 10: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Week 12; Test type: Superiority or Other; p = 0.5474, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 36.0, 90% CI 2-sided [-62.44 to 134.38]
Statistical Analysis 11: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo,Week 12; Test type: Superiority or Other; p = 0.1918, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 78.5, 90% CI 2-sided [-20.48 to 177.56]
Statistical Analysis 12: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Week 12; Test type: Superiority or Other; p = 0.9615, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -3.0, 90% CI 2-sided [-104.88 to 98.91]

9. Secondary Outcome: Percent Change From Baseline in High Sensitivity C-reactive Protein (hsCRP) at Weeks 4, 8, and 12
Description: hsCRP was one of the PD biomarkers of the study.
Time Frame: Baseline; Weeks 4, 8, and 12
Population: as for outcome 8
Measure: Geometric Mean (90% Confidence Interval); unit: percent change
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 73 | 71 | 72 | 71 | 70
percent change
  Week 4 (n=67,64,69,71,65) | -11.60 [-25.69 to 5.17] | -19.17 [-34.22 to -0.67] | -26.90 [-39.41 to -11.82] | -35.21 [-49.10 to -17.55] | -17.70 [-30.08 to -3.13]
  Week 8 (n=71,63,69,71,68) | -2.42 [-22.75 to 23.25] | -6.00 [-23.09 to 14.89] | -31.43 [-44.11 to -15.88] | -43.15 [-54.57 to -28.86] | -22.70 [-36.72 to -5.59]
  Week 12 (n=67,62,68,71,64) | 14.85 [-11.16 to 48.48] | 4.51 [-18.02 to 33.25] | -20.40 [-38.61 to 3.22] | -15.96 [-33.12 to 5.60] | 2.31 [-18.48 to 28.42]
Statistical Analysis 1: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Week 4; Test type: Superiority or Other; p = 0.9328, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 6.4, 90% CI 2-sided [-118.60 to 131.41]
Statistical Analysis 2: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Week 4; Test type: Superiority or Other; p = 0.8962, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -9.8, 90% CI 2-sided [-132.91 to 113.39]
Statistical Analysis 3: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, Week 4; Test type: Superiority or Other; p = 0.8775, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 11.5, 90% CI 2-sided [-110.83 to 133.74]
Statistical Analysis 4: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Week 4; Test type: Superiority or Other; p = 0.8224, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -17.0, 90% CI 2-sided [-142.02 to 107.94]
Statistical Analysis 5: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Week 8; Test type: Superiority or Other; p = 0.4831, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -52.7, 90% CI 2-sided [-176.48 to 71.02]
Statistical Analysis 6: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Week 8; Test type: Superiority or Other; p = 0.1183, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -115.2, 90% CI 2-sided [-236.63 to 6.13]
Statistical Analysis 7: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, Week 8; Test type: Superiority or Other; p = 0.1139, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -115.8, 90% CI 2-sided [-236.29 to 4.69]
Statistical Analysis 8: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Week 8; Test type: Superiority or Other; p = 0.1931, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -96.4, 90% CI 2-sided [-218.17 to 25.46]
Statistical Analysis 9: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, Week 12; Test type: Superiority or Other; p = 0.1182, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -119.7, 90% CI 2-sided [-245.66 to 6.32]
Statistical Analysis 10: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, Week 12; Test type: Superiority or Other; p = 0.5784, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -41.7, 90% CI 2-sided [-165.34 to 81.87]
Statistical Analysis 11: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo,Week 12; Test type: Superiority or Other; p = 0.0279, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -163.6, 90% CI 2-sided [-285.84 to -41.29]
Statistical Analysis 12: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, Week 12; Test type: Superiority or Other; p = 0.1053, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -123.5, 90% CI 2-sided [-249.00 to 1.93]

10. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score at Week 12
Description: IBDQ: Psychometrically validated patient reported outcome (PRO) instrument for measuring disease-specific quality of life (QOL) in participants with inflammatory bowel disease. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). Total score is the sum of each item score, ranged from 32 to 224 with higher score indicating better QOL. Positive change in total score indicated improvement in QOL.
Time Frame: Baseline, Week 12
Population: The primary analysis population was based on an mITT analysis set, which was defined as all randomized participants who received at least 1 dose of randomized treatment. n=number of evaluable participants at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 73 | 71 | 72 | 71 | 70
units on a scale
  Baseline (BL)(n=69,68,65,71,66) | 128.0 (30.69) [-2.043 to -1.014] | 122.1 (38.82) [-2.944 to -1.881] | 133.4 (34.79) [-3.570 to -2.550] | 128.0 (32.42) [-3.162 to -2.131] | 132.3 (36.84) [-3.337 to -2.270]
  Change at W12 (n=62,55,61,64,54) | 19.8 (34.08) [-2.280 to -1.171] | 20.1 (35.24) [-3.241 to -2.084] | 32.7 (34.10) [-3.866 to -2.775] | 32.1 (31.70) [-3.357 to -2.236] | 36.2 (29.45) [-3.583 to -2.442]
Statistical Analysis 1: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, change from BL at W12; Test type: Superiority or Other; p = 0.8302, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -1.10, 90% CI 2-sided [-9.507 to 7.317]
Statistical Analysis 2: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, change from BL at W12; Test type: Superiority or Other; p = 0.0141, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 12.33, 90% CI 2-sided [4.084 to 20.567]
Statistical Analysis 3: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, change from BL at W12; Test type: Superiority or Other; p = 0.0182, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 11.70, 90% CI 2-sided [3.564 to 19.840]
Statistical Analysis 4: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, change from BL at W12; Test type: Superiority or Other; p = 0.0026, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 15.48, 90% CI 2-sided [7.056 to 23.907]

11. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Domain Scores at Week 12
Description: IBDQ: Psychometrically validated PRO instrument for measuring disease-specific QOL in participants with inflammatory bowel disease. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). Total score is the sum of each item score, ranged from 32 to 224 with higher score indicating better QOL. Positive change in total score indicated improvement in QOL. There are 4 individual domains under the IBDQ: bowel function (fx)/symptoms (score range of 10-70), systemic symptoms (score range of 5-35), emotional status/fx (score range of 12-84), and social fx (score range of 5-35). As with total score, higher scores indicate better QOL in that domain.
Time Frame: Baseline (BL), Week 12
Population: The primary analysis population was based on an mITT analysis set, which was defined as all randomized participants who received at least 1 dose of randomized treatment. n=number of evaluable participants at the specified time point for that specific domain.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 73 | 71 | 72 | 71 | 70
units on a scale
  BL, bowel fx (n=69,68,65,71,66) | 38.9 (9.96) [-2.043 to -1.014] | 37.0 (12.23) [-2.944 to -1.881] | 41.7 (10.60) [-3.570 to -2.550] | 38.5 (9.95) [-3.162 to -2.131] | 41.0 (11.37) [-3.337 to -2.270]
  Change at W12, bowel fx (n=62,55,61,64,54) | 7.4 (11.93) [-2.280 to -1.171] | 6.9 (12.51) [-3.241 to -2.084] | 11.3 (11.05) [-3.866 to -2.775] | 11.8 (12.07) [-3.357 to -2.236] | 12.8 (11.45) [-3.583 to -2.442]
  BL, emotional fx (n=69,68,65,71,66) | 50.4 (12.60) | 48.4 (15.39) | 51.2 (14.70) | 50.4 (13.73) | 51.3 (15.92)
  Change at W12, emotional fx (n=62,55,61,64,54) | 5.9 (11.91) | 6.6 (12.22) | 10.8 (13.85) | 10.0 (12.04) | 12.0 (11.40)
  BL, systemic symptoms (SS)(n=69,68,65,71,66) | 18.1 (5.62) | 18.2 (6.81) | 19.6 (5.98) | 18.4 (6.42) | 19.0 (5.97)
  Change at W12, SS (n=62,55,61,64,54) | 3.3 (6.67) | 3.1 (5.95) | 4.7 (5.91) | 4.9 (5.49) | 4.8 (5.05)
  BL, social fx (n=69,68,65,71,66) | 20.6 (7.87) | 18.5 (8.07) | 20.9 (7.37) | 20.7 (6.99) | 20.9 (7.73)
  Change at W12, social fx (n=62,55,61,64,54) | 3.3 (6.27) | 3.6 (7.33) | 5.9 (6.51) | 5.4 (6.90) | 6.6 (6.58)
Statistical Analysis 1: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, bowel fx change from BL at W12; Test type: Superiority or Other; p = 0.6862, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.73, 90% CI 2-sided [-3.689 to 2.235]
Statistical Analysis 2: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, bowel fx change from BL at W12; Test type: Superiority or Other; p = 0.0135, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 4.37, 90% CI 2-sided [1.467 to 7.280]
Statistical Analysis 3: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, bowel fx change from BL at W12; Test type: Superiority or Other; p = 0.0171, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 4.16, 90% CI 2-sided [1.293 to 7.023]
Statistical Analysis 4: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, bowel fx change from BL at W12; Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 5.20, 90% CI 2-sided [2.232 to 8.172]
Statistical Analysis 5: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, emotional fx change from BL at W12; Test type: Superiority or Other; p = 0.9072, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 0.22, 90% CI 2-sided [-2.897 to 3.339]
Statistical Analysis 6: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, emotional fx change from BL at W12; Test type: Superiority or Other; p = 0.0161, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 4.47, 90% CI 2-sided [1.420 to 7.522]
Statistical Analysis 7: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, emotional fx change from BL at W12; Test type: Superiority or Other; p = 0.0271, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 4.06, 90% CI 2-sided [1.042 to 7.071]
Statistical Analysis 8: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, emotional fx change from BL at W12; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 5.90, 90% CI 2-sided [2.778 to 9.026]
Statistical Analysis 9: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, systemic symptoms change from BL at W12; Test type: Superiority or Other; p = 0.7711, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.26, 90% CI 2-sided [-1.756 to 1.229]
Statistical Analysis 10: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, systemic symptoms change from BL at W12; Test type: Superiority or Other; p = 0.0582, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 1.69, 90% CI 2-sided [0.223 to 3.147]
Statistical Analysis 11: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, systemic symptoms change from BL at W12; Test type: Superiority or Other; p = 0.0558, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 1.68, 90% CI 2-sided [0.235 to 3.120]
Statistical Analysis 12: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, systemic symptoms change from BL at W12; Test type: Superiority or Other; p = 0.0686, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 1.66, 90% CI 2-sided [0.161 to 3.153]
Statistical Analysis 13: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo, social fx change from BL at W12; Test type: Superiority or Other; p = 0.7561, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = -0.33, 90% CI 2-sided [-2.094 to 1.429]
Statistical Analysis 14: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo, social fx change from BL at W12; Test type: Superiority or Other; p = 0.0384, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 2.17, 90% CI 2-sided [0.447 to 3.891]
Statistical Analysis 15: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo, social fx change from BL at W12; Test type: Superiority or Other; p = 0.0729, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 1.86, 90% CI 2-sided [0.154 to 3.557]
Statistical Analysis 16: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo, social fx change from BL at W12; Test type: Superiority or Other; p = 0.0060, Mixed Models Analysis; [statistical method as in outcome 6, analysis 2]; LSM Difference = 2.95, 90% CI 2-sided [1.190 to 4.715]

12. Secondary Outcome: Percentage of Participants With an Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score of More Than or Equal to (>=) 170 at Week 12
Description: IBDQ: Psychometrically validated PRO instrument for measuring disease-specific QOL in participants with inflammatory bowel disease. IBDQ consists of 32 items, each item score ranged from 1 (worst possible response) to 7 (best possible response). Total score is sum of each item score, ranged from 32 to 224 with higher score indicating better QOL. Positive change in total score indicated improvement in QOL. A score of >=170 corresponds to clinical remission.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 65 | 57 | 63 | 64 | 54
percentage of participants | 36.9 [27.4 to 47.5] | 36.8 [26.9 to 47.9] | 55.6 [45.0 to 66.3] | 46.9 [36.1 to 57.5] | 48.1 [36.3 to 59.4]
Statistical Analysis 1: Comparison: Placebo vs PF-00547659 7.5 mg; PF-00547659 7.5 mg vs placebo; Test type: Superiority or Other; p = 0.5201, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = -0.002, 90% CI 2-sided [-0.145 to 0.142] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 2: Comparison: Placebo vs PF-00547659 22.5 mg; PF-00547659 22.5 mg vs placebo; Test type: Superiority or Other; p = 0.0217, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.183, 90% CI 2-sided [0.039 to 0.328] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 3: Comparison: Placebo vs PF-00547659 75 mg; PF-00547659 75 mg vs placebo; Test type: Superiority or Other; p = 0.1473, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.096, 90% CI 2-sided [-0.045 to 0.237] — Statistics of risk difference are calculated using the Minimum Risk Weights test
Statistical Analysis 4: Comparison: Placebo vs PF-00547659 225 mg; PF-00547659 225 mg vs placebo; Test type: Superiority or Other; p = 0.1231, Cochran-Mantel-Haenszel — 1-sided p-value; Statistics of risk difference are calculated using the Minimum Risk Weights test; Risk Difference (RD) = 0.112, 90% CI 2-sided [-0.038 to 0.261] — Statistics of risk difference are calculated using the Minimum Risk Weights test

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Withdrawals Due to TEAEs During the Treatment Period (Weeks 0-12)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. TEAEs are defined as newly occurring AEs or those worsening after first dose. AEs comprised both SAEs and non-SAEs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Screening through to end of treatment period, up to 12 weeks
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 73 | 71 | 70 | 73 | 70
participants
  With TEAEs | 39 | 41 | 36 | 43 | 43
  With SAEs | 4 | 11 | 1 | 3 | 3
  Withdrawals due to TEAEs | 2 | 5 | 0 | 3 | 1

14. Secondary Outcome: Maximum Serum PF-00547659 Concentration Achieved
Time Frame: Weeks 0 (baseline), 2, 4,8, 12, 16, 20, 24, 28, 32, and 36; Early Withdrawal
Population: Participants who received active treatment (PF-00547659) were included in this analysis.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Number analyzed (Participants) | 0 | 67 | 67 | 68 | 62
nanograms (ng)/milliliter (mL) |  | 929.4 (1977.8) | 2062 (1395.5) | 6576 (2146.0) | 21470 (4788.4)

ADVERSE EVENTS:
Time Frame: Screening till Week 36 or Early Withdrawal, whichever was later.
Description: Two subjects initially randomized to the 22.5 mg group were mistakenly administered the 75 mg dose instead.
Arm/Group | Placebo | PF-00547659 7.5 mg | PF-00547659 22.5 mg | PF-00547659 75 mg | PF-00547659 225 mg
Serious Adverse Events (participants affected / at risk) | 4/73 | 11/71 | 2/70 | 4/73 | 3/70
Other Adverse Events (participants affected / at risk) | 17/73 | 16/71 | 15/70 | 14/73 | 18/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | PF-00547659 7.5 mg (N=71) | PF-00547659 22.5 mg (N=70) | PF-00547659 75 mg (N=73) | PF-00547659 225 mg (N=70)
Retinal artery embolism (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 6 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Colectomy total (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | PF-00547659 7.5 mg (N=71) | PF-00547659 22.5 mg (N=70) | PF-00547659 75 mg (N=73) | PF-00547659 225 mg (N=70)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 6 | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 6 | 1 | 1 | 4
Vomiting (Gastrointestinal disorders) | 3 | 1 | 4 | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 0 | 3 | 5 | 4
Headache (Nervous system disorders) | 6 | 5 | 7 | 4 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.